CLINICAL TRIAL: NCT04493229
Title: A Pilot Feasibility Study of Intramuscular Oxytocin on Fear of Pain and Trust in Physical Therapist During Outpatient Rehabilitation After Total Knee Arthroplasty
Brief Title: A Pilot Feasibility Study of IM OXT on Fear of Pain and Trust in Physical Therapist During OP Rehabilitation After TKA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study team decided not to proceed with project
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00066646
Record Dates: First submitted 2020-07-16; First posted 2020-07-30 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2020-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind study of oxytocin (IM) or placebo given
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oxytocin (Experimental): Oxytocin IM injection will be given per randomization prior to first outpatient physical therapy session
  Interventions: Drug: Oxytocin
- Placebo (Active Comparator): Placebo IM injection will be given per randomization prior to first outpatient physical therapy session
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — IM Oxytocin
  Other Names: Pitocin
  Arms: Oxytocin
Drug: Placebo — Placebo IM
  Arms: Placebo

SUMMARY:
This study will examine the effect that a dose of intramuscular (IM) oxytocin (naturally occurring hormone) has on fear of pain and movement and trust in the physical therapist during outpatient rehabilitation after total knee replacement has been performed. Investigators will ask participants to answer questions about fear of pain and movement before several outpatient physical therapy session and investigators will ask participants questions about trust of the physical therapist several times after the outpatient physical therapy sessions.

DETAILED DESCRIPTION:
The purpose of this study is to determine feasibility of this study design and identify barriers that altered design could bring to overcome these barriers in the design of a large, pragmatic, multi-center clinical trial. It is also designed to estimate the effect size and variance of the main outcome measures, trust and fear, in patients undergoing rehabilitation after total knee arthroplasty (TKA). The study team hypothesizes that intramuscular (IM) oxytocin, in a dose and time determined by a series of previous studies under this grant to target the brain, will enhance trust and reduce fear and that these will be associated with improved outcomes. Again, the study is not designed to test this hypothesis, but to gather the critical data necessary to test it in a large, multi-center clinical trial that would follow this grant.

Participants that have decided to undergo unilateral TKA, will come to the Pain Clinical Research Unit at least 48 hours prior to surgery to confirm consent and complete a series of questionnaires. Participants surgery, anesthesia, and postoperative medication and therapy treatment will be routine. On the first outpatient study visit participants will complete a questionnaire of fear about pain and receive an intramuscular injection of oxytocin or placebo in a randomized, double blind manner. At the end of this session participants will complete a questionnaire assessing the degree of trust in the therapist. Physical therapy be will routine, and the fear and trust questionnaires will be completed at the 2nd, 4th, 8th, and last physical therapy session as well as routine measures of progress and function. The primary outcome measure is assessment of effect size and variability of the trust and fear questionnaires on the 1st and 2nd visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 and < 75 years of age, Body Mass Index (BMI) <40.
2. Generally in good health as determined by the Principal Investigator based on prior medical history, American Society of Anesthesiologists physical status 1, 2, or 3. Scheduled for unilateral TKA and postoperative physical therapy at Davie Medical Center.
3. Normal blood pressure (systolic 90-140 mmHg; diastolic 50-90 mmHg) resting heart rate 45-100 beats per minute) without medication or for those with hypertension, pressure controlled with anti-hypertensives and with a resting heart rate 45-100 beats per minute.
4. Female subjects of child-bearing potential and those < 1 year post-menopausal, must be practicing highly effective methods of birth control such as hormonal methods (e.g., combined oral, implantable, injectable, or transdermal contraceptives), double barrier methods (e.g., condoms, sponge, diaphragm, or vaginal ring plus spermicidal jellies or cream), or total abstinence from heterosexual intercourse for a minimum of 1 full cycle before study drug administration.

Exclusion Criteria:

1. Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
2. Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (active gynecologic disease in which increased tone would be detrimental e.g., uterine fibroids with ongoing bleeding), compromise the subject's compliance with study procedures, or compromise the quality of the data
3. Women who are pregnant (positive result for urine pregnancy test at screening visit), women who are currently nursing or lactating, women that have been pregnant within 2 years
4. Subjects with neuropathy, chronic pain, diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Tampa Scale of Kinesiophobia-11 (TSK-11) | Postoperative Outpatient Physical Therapy Visit 1/study medication administration visit/Baseline
  TSK-11 scale ranges from 11 to 44 with a higher score denoting a worse outcome.
  The TSK-11 will be completed prior to the outpatient post-operative physical therapy session
Tampa Scale of Kinesiophobia-11 (TSK-11) | Postoperative Outpatient Physical Therapy Visit 2, 1-5 days after study medication
  TSK-11 scale ranges from 11 to 44 with a higher score denoting a worse outcome.
  The TSK-11 will be completed prior to the outpatient post-operative physical therapy session
Tampa Scale of Kinesiophobia-11 (TSK-11) | Postoperative Outpatient Physical Therapy Visit 4, 5-10 days after study medication
  TSK-11 scale ranges from 11 to 44 with a higher score denoting a worse outcome.
  The TSK-11 will be completed prior to the outpatient post-operative physical therapy session
Tampa Scale of Kinesiophobia-11 (TSK-11) | Postoperative Outpatient Physical Therapy Visit 8, 7 -20 days after study medication
  TSK-11 scale ranges from 11 to 44 with a higher score denoting a worse outcome.
  The TSK-11 will be completed prior to the outpatient post-operative physical therapy session
Tampa Scale of Kinesiophobia-11 (TSK-11) | Postoperative Outpatient Physical Therapy Final Visit, 10-60 days after study medication
  TSK-11 scale ranges from 11 to 44 with a higher score denoting a worse outcome.
  The TSK-11 will be completed prior to the outpatient post-operative physical therapy session
Working Alliance Inventory (WAI) | Postoperative Outpatient Physical Therapy Visit 1/study medication administration visit/Baseline
  The WAI score ranges from 24 to 72 with a higher score denoting a better outcome.
  The WAI will be completed after the outpatient post-operative physical therapy session.
Working Alliance Inventory (WAI) | Postoperative Outpatient Physical Therapy Visit 2, 1-5 days after study medication
  The WAI score ranges from 24 to 72 with a higher score denoting a better outcome.
  The WAI will be completed after the outpatient post-operative physical therapy session.
Working Alliance Inventory (WAI) | Postoperative Outpatient Physical Therapy Visit 4, 5-10 days after study medication
  The WAI score ranges from 24 to 72 with a higher score denoting a better outcome.
  The WAI will be completed after the outpatient post-operative physical therapy session.
Working Alliance Inventory (WAI) | Postoperative Outpatient Physical Therapy Visit 8, 7 -20 days after study medication
  The WAI score ranges from 24 to 72 with a higher score denoting a better outcome.
  The WAI will be completed after the outpatient post-operative physical therapy session.
Working Alliance Inventory (WAI) | Postoperative Outpatient Physical Therapy Final Visit, 10-60 days after study medication
  The WAI score ranges from 24 to 72 with a higher score denoting a better outcome.
  The WAI will be completed after the outpatient post-operative physical therapy session.

SECONDARY OUTCOMES:
Pain during straight leg raise | Post-operative outpatient physical therapy sessions, up to 12 weeks post surgery
  During the postoperative physical therapy sessions, pain using a 0-10 verbal scale, with 0 equivalent to NO PAIN and 10 equivalent to THE WORST PAIN IMAGINABLE will be measured and the data collected from the electronic medical record.
Pain after straight leg raise | Post-operative outpatient physical therapy sessions, up to 12 weeks post surgery
  During the postoperative physical therapy sessions, pain using a 0-10 verbal scale, with 0 equivalent to NO PAIN and 10 equivalent to THE WORST PAIN IMAGINABLE will be measured and the data collected from the electronic medical record.
Physical therapist deems stepping exercise begins; may walk up and down steps | Post-operative 24-48 hours after surgery
  During routine physical therapy after this surgery, the therapist determines when the patient is ready to begin stepping exercised during therapy. It is a subjective determination by the therapist. The outcome measure is the number of days since surgery when the therapist notes in the electronic medical record (EMR) that the patient began stepping exercises.
Gait speed | Post-operative outpatient physical therapy sessions, up to 12 weeks post surgery
  Gait speed will be measured by the physical therapist at the first physical therapy session and the last physical therapy session and at varying times during physical therapy after surgery using meters/seconds. Distance in meters is divided by the number of seconds.
  This data will be recorded in the electronic medical recorded and recorded from the electronic medical record.
Average pain score | Post-operative outpatient physical therapy sessions, up to 12 weeks post surgery
  Patients will be asked to verbally state the average pain they have experienced in the 24 hours prior to the scheduled physical therapy session. Average pain will be measured using a verbal pain scale; 0 is equivalent to NO PAIN and 10 is equivalent to THE WORST PAIN IMAGINABLE.
Analgesic Consumption | Post-operative outpatient physical therapy sessions, up to 12 weeks post surgery
  Analgesic medications will be recorded from the day previous to each therapy session. Analgesic consumption will be converted into morphine equivalents using a standard conversion table.

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No